CLINICAL TRIAL: NCT05485974
Title: A Phase 1, Open Label, Dose Escalation of HBI-2438 in Patients With Advanced Malignant Solid Tumors Harboring KRAS G12C Mutation
Brief Title: A Dose Escalation Study of HBI-2438 in Patients With Solid Tumors Harboring KRAS G12C Mutation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBI-2438-101
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Colorectal Cancer; Cancer of Pancreas; Colon Cancer; Solid Tumor; Cancer
Keywords: KRAS G12C; FIH
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation Design with Expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): HBI-2438 will be given orally in ascending doses (escalation cohort), until the maximum tolerated dose or recommended Phase 2 dose is reached. Up to 6-8 patients will then be enrolled in the expansion cohort at the recommended dose.
  Interventions: Drug: HBI-2438

INTERVENTIONS:
Drug: HBI-2438 — KRAS G12C Inhibitor

SUMMARY:
A Phase 1 dose escalation study in patients with advanced solid tumors harboring KRAS G12C mutation to determine the maximum tolerated dose and recommended Phase II dose of HBI-2438 and characterize its pharmacokinetic profile.

DETAILED DESCRIPTION:
A Phase 1, Open-Label, Dose Escalation of HBI-2438 in Patients with Advanced Malignant Solid Tumors Harboring KRAS G12C Mutation. The primary and secondary objectives are:

1. To determine the MTD and recommended Phase 2 dose (RP2D) of HBI-2438 as an oral monotherapy for advanced solid tumors harboring KRAS G12C mutation.
2. To characterize the PK of HBI-2438 in subjects with advanced malignant solid tumors harboring KRAS G12C mutation.

HBI-2438 is an orally administered KRAS G12C Inhibitor and will be dosed once daily throughout the escalation and expansion phase. Up to 44 subjects will be enrolled sequentially into the 3+3 dose escalation and monitored throughout the study for safety and tolerability. The dose escalation phase will consist of 6 cohorts, with doses ranging from 150 to 1200mg. Once the MTD of RP2D is established, an additional 6-8 subjects with brain metastases will be enrolled into the expansion phase at that dose level.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

Male or female at least 18 years of age at the time of signing the ICF prior to initiation of any study specific activities/procedures

Advanced malignant solid tumors with KRAS G12C mutation- as determined by genetic testing

Must have failed or refused standard of care therapy, are not eligible for standard of care therapy, or cannot benefit from standard of care therapy, in the opinion of the Investigator

At least 1 measurable target lesion that meets the definition of RECIST v1.1

ECOG Performance Status of 0 or 1

Demonstrate adequate organ function

Expected survival time > 3 months in the opinion of the investigator

Must be able to swallow oral medications and must not have gastrointestinal abnormalities that significantly affect drug absorption

Exclusion Criteria:

Key Exclusion Criteria:

History of another concurrent malignancy within 3 years prior to study entry, unless the malignancy was treated with curative intent and the likelihood of relapse is <5% in 2 years Note: Subjects with a history of squamous or basal cell carcinoma of the skin or carcinoma in the situ of the cervix may be enrolled

Untreated or symptomatic central nervous system (CNS) metastases Note: Subjects with asymptomatic treated CNS metastases are eligible provided they have been clinically stable and not requiring steroids for at least 4 weeks

Clinically significant cardiovascular disease, including stroke or myocardial infarction within 6 months prior to first dose of HBI-2438; or the presence of unstable angina or congestive heart failure of New York Heart Association Grade 2 or higher

Any unresolved Grade 2 or greater toxicity from previous anti-cancer therapy, except alopecia, within 4 weeks of first study treatment administration

Active autoimmune diseases or history of autoimmune diseases that may relapse

Pregnant or nursing

Prior treatment with any KRAS G12C inhibitors

Any condition that required systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤14 days before the first study treatment administration

Treatment with other investigational drugs/devices within 4 weeks prior to first study treatment administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) | Up to 36 months
  Safety endpoints: Incidence of dose-limiting toxicities (DLTs)
adverse events (AEs), and serious adverse events (SAEs) overall | Up to 36 months
  Safety endpoints: adverse events (AEs), and serious adverse events (SAEs) overall

SECONDARY OUTCOMES:
maximum plasma concentration (Cmax) | Cycle 1 (21 days)
  Pharmacokinetic variables including maximum plasma concentration (Cmax)
minimum plasma concentration (Cmin) | Cycle 1 (21 days)
  Pharmacokinetic variables including minimum plasma concentration (Cmin)
Area Under the Curve (AUC) | Cycle 1 (21 days)
  Pharmacokinetic variables including Area Under the Curve (AUC)
Pharmacokinetic variables including clearance | Cycle 1 (21 days)
  Pharmacokinetic variables including clearance
Pharmacokinetic variables including serum half-life | Cycle 1 (21 days)
  Pharmacokinetic variables including serum half-life
Pharmacokinetic variables including volume of distribution | Cycle 1 (21 days)
  Pharmacokinetic variables including volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Bessudo, MD, Principal Investigator — California Cancer Associates for Research and Excellence, Inc. (cCare)
Locations (14):
- United States (13):
  - California Cancer Associates for Research and Excellence, Inc. (cCare), Encinitas, California
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - The Oncology Institute of Hope and Innovation, Long Beach, California
  - The Oncology Institute of Hope and Innovation, Pasadena, California
  - California Cancer Associates for Research and Excellence, Inc. (cCare), San Marcos, California
  - The Oncology Institute of Hope and Innovation, Santa Ana, California
  - Sarcoma Oncology, Santa Monica, California
  - Innovative Clinical Research Institute (ICRI), Whittier, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - BRCR Medical Center, Plantation, Florida
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Gabrail Cancer Center, Canton, Ohio
- Pan American Center for Oncology Trials (PanOncology Trials), Rio Piedras, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No